CLINICAL TRIAL: NCT06962917
Title: Examining the Network Structure of Social Anxiety and Body Dysmorphic Symptoms in American, German, and Japanese: A Cross-Cultural Study
Brief Title: Cross-Cultural Differences in the Network Structure of Social Anxiety and Body Dysmorphic Symptoms
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01k-rev
Record Dates: First submitted 2025-03-28; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Depression; Anxiety; Body Dysmorphic Disorders
Keywords: Cross-cultural study
MeSH Terms: conditions — Depression; Anxiety Disorders; Body Dysmorphic Disorders | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- German, American, and Japanese citizens over 18 years old
  Interventions: Other: Cross sectional study

INTERVENTIONS:
Other: Cross sectional study — This study is a cross-cultural study, not an intervention study. A total of 1,523 participants (484 from Germany, 548 from the United States, and 491 from Japan) were recruited.

SUMMARY:
This study will examine cross-cultural differences in the network structure of social anxiety and body dysmorphic symptoms across Germany, the United States, and Japan.

DETAILED DESCRIPTION:
This study will investigate the network structure of social anxiety, body dysmorphic symptoms, depressive symptoms, and shame across Germany, the United States, and Japan. Social anxiety disorder and body dysmorphic disorder frequently co-occur and share several clinical features beyond fear of negative evaluation (Coles et al., 2006; Dietel et al., 2021; Fang et al., 2011). Both conditions have also been found to exhibit high comorbidity with major depressive disorder (Acarturk et al., 2008; Grant et al., 2005; Gunstad & Phillips, 2003; Phillips et al., 1998). Cognitive-behavioral therapy targeting social anxiety disorder or body dysmorphic disorder has been shown to significantly alleviate depressive symptoms (e.g., Enander et al., 2016; Noda et al., 2023; Ritter et al., 2023). Shame has also been implicated in the development of depressive symptoms, as well as social anxiety disorder and body dysmorphic disorder (Kim et al., 2011). Comparing the symptom networks of social anxiety, body dysmorphic symptoms, and depression-and identifying central symptoms within each cultural context-may contribute to the development of transdiagnostic treatments with cross-cultural applicability.

ELIGIBILITY:
Inclusion Criteria:

* German, American, and Japanese citizens over 18 years old.

Exclusion Criteria:

* Individuals who do not obtain consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: German, American, and Japanese individuals
Sampling Method: Probability Sample
Enrollment: 1523 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Brief version of Fear of Negative Evaluation scale | From March 2025 to April 2025
  The Brief version of Fear of Negative Evaluation scale measures fear of negative evaluation. The scale consists of 12 items, including eight for the straightforwardly worded items and four for the reverse worded items. Each item is rated on a 5-point scale ranging from 1 (not characteristic of me) to 5 (extremely characteristic of me), with higher scores indicating greater fear of negative evaluation. It is recommended that the straightforwardly worded items (8 items) are used for the assessment of fear of negative evaluation. The total score, based on all 12 items, ranges from 12 to 60. When using only the straightforwardly worded items, the total score ranges from 8 to 40.
Mini-Social Phobia Inventory | From March 2025 to April 2025
  The Mini-social phobia inventory measures social anxiety and avoidance behavior. The scale contains three items rated on a 5-point scale from 0 (not at all) to 4 (extremely), with higher scores indicating greater social anxiety symptoms. The total score ranges from 0 to 12.
Appearance Anxiety Inventory. | From March 2025 to April 2025
  The Appearance Anxiety Inventory measures symptoms of body dysmorphic disorder. The scale contains ten items rated on a 5-point scale from 0 (not at all) to 4 (all the time), with higher scores indicating greater symptoms of body dysmorphic disorder. The total score ranges from 0 to 40, with scores of 19 or above indicating caseness.
Patient Health Questionnaire-9 | From March 2025 to April 2025
  The Patient Health Questionnaire-9 assesses depressive symptoms. It consists of nine items, each rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day), with higher scores indicating more severe depressive symptoms. The total score ranges from 0 to 27.
External and Internal Shame Scale | From March 2025 to April 2025
  The External and Internal Shame Scale measures external shame and internal shame. It consists of eight items, each rated on a 5-point scale ranging from 0 (never) to 4 (always), with higher scores indicating greater levels of shame. The total score ranges from 0 to 32.
Auckland individualism and collectivism scale | From March 2025 to April 2025
  The Auckland individualism and collectivism scale measures individualism (competitiveness, uniqueness, and responsibility) and collectivism (advise and harmony). The scale consists of 26 items, each rated on a 6-point scale ranging from 1 (never or almost never) to 6 (always), with higher scores indicating greater levels of the respective construct. The total score ranges from 26 to 156.
Demographic data | From March 2025 to April 2025
  Age, location, ethnicity, education history, sexual orientation, biological sex, Gender identity, etc.

OTHER OUTCOMES:
LGBTQIA+ minority stress questionnaire | From March 2025 to April 2025
  The LGBTQIA+ minority stress questionnaire measures level of stress of LGBTQIA+ minority. The scale contains 19 items rated on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree), with higher scores indicating greater level of stress of LGBTQIA+ minority. The total score ranges from 0 to 76.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Marburg, Hesse, Germany